## Study Title: Intervention to Educate and Improve Underserved Population's Uptake and Completion of the HPV Vaccine Series

**Principal Investigator: Evelinn Borrayo** 

COMIRB No: 19-2236 Version Date: 2/19/2025

You are being asked to be in this research study because you are either a parent of an adolescent (9-17-year-old) or are a young adult 18-26 years old and are interested in knowing more about the HPV vaccine.

If you join the study, you will be asked to participate in an educational session regarding HPV related cancers and the HPV vaccine. The educational materials could be presented in person or sent to you via email, text, or through MyChart in your Denver Health electronic health record. You will complete a 5-minute survey after watching educational materials and will receive a \$25 gift card after completing the survey.

Additionally, if you agree to be in the study, the CU Cancer Center staff will access your personal health information (PHI) at Denver Health to help you obtain a dose of the HPV vaccine. PHI will be accessed using your medical record number or the medical record of your participating child to verify HPV vaccination status via your Epic chart (electronic health record) and the Colorado Immunization Information System (CIIS) If you choose to obtain the vaccine, a patient navigator or scheduler will schedule a vaccine administration at your primary care clinic

This study is designed to learn more about your thoughts and beliefs about HPV related cancers, as well as how HPV education and patient navigation help improve HPV vaccination rates.

Possible discomforts or risks include feeling uncomfortable answering personal questions. There may be risks the researchers have not thought of.

Every effort will be made to protect your privacy and confidentiality by storing records using electronic data sources which are password-protected and available only to the study team.

You have a choice about being in this study. You do not have to be in this study if you do not want to be.

The data we collect will be used for this study but may also be important for future research. Your unidentified data may be used for future research or distributed to other researchers for future study without additional consent, but the information that identifies you will be removed from the data.

If you have questions, you can call Mona Krull, at 303-602-9716. You can call and ask questions at any time.

You may have questions about your rights as someone in this study. If you have questions, you can call the COMIRB (the responsible Institutional Review Board). Their number is (303) 724-1055.

By completing the survey, you are agreeing to participate in this research study.

Postcard Consent CF-157, Effective 4-26-2010